CLINICAL TRIAL: NCT00314665
Title: Use of Thalidomide in Chronic Uveitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-08-28-05
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Uveitis
Keywords: Sarcoidosis; Chronic Uveitis; Uveitis; Thalidomide
MeSH Terms: conditions — Uveitis; Sarcoidosis | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
This research study is for patients that have been diagnosed with chronic uveitis, a disease that causes inflammation in the eye. Patients are currently being treated with Remicade, Humira, Methotrexate and or similar chemotherapy type drugs to control this inflammation. Despite these medications, patients still have inflammation in their eyes. Patients are being asked to add an additional drug, thalidomide.

DETAILED DESCRIPTION:
Patients will be in the study for approximately 24 weeks. The visits are at screening, baseline (week 0), and weeks 4,8,12, and 24.

The purpose of this research study is to see if Thalidomide is safe and effective in the treatment of patients with chronic inflammation in their eyes. Thalidomide is approved by the Food and Drug Administration (FDA) for a leprosy skin condition, erythema nodosum leprosum (ENL). The drug works in many different ways, including as an anti-inflammation drug. Therefore, it is thought that this drug might be able to improve symptoms and lung function. At this time, the drug is not approved for use for uveitis.

ELIGIBILITY:
Inclusion Criteria:

* You are being asked to take part in this research study because you have been diagnosed with chronic uveitis, a disease that causes inflammation in the eye. You are currently being treated with Remicade, Humira, Methotrexate and or similar chemotherapy type drugs to control this inflammation. Despite these medications, you still have inflammation in your eyes. You are being asked to add an additional drug, thalidomide.

Exclusion Criteria:

* You will not participate in this research study if any of the following apply to you:

  * Pregnant
  * If you are a man or woman not willing to take adequate birth control measures comply with FDA-mandated S.T.E.P.S.â program. .
  * If you are a breast feeding woman
  * If you have a significant peripheral neuropathy (numbness or tingling in your hands or feet)
  * Have had a recent blood clot in your leg or lungs
  * If you are currently receiving biphosphonates such as zoledronic acid (fosamax)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2004-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Need for corticosteroids to control eyes
Global assessment of ocular status

SECONDARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Principal Investigator — Professor of Medicine
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States